CLINICAL TRIAL: NCT04869670
Title: A Pilot and Feasibility Trial of G-POEM for Gastroparesis to Assess Safety, Physiological Mechanisms and Efficacy
Brief Title: A Study to Evaluate Safety and Effectiveness of G-POEM for Gastroparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Johns Hopkins University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-001928; R01DK125680 (NIH)
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Gastroparesis
Keywords: Gastric Peroral Endoscopic Pyloromyotomy (G-POEM)
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-POEM (Experimental)
  Interventions: Procedure: Gastric peroral endoscopic myotomy.
- Sham procedure (Sham Comparator)
  Interventions: Procedure: Sham Gastric peroral endoscopic myotomy.

INTERVENTIONS:
Procedure: Gastric peroral endoscopic myotomy. — Under propofol anesthesia, EndoFLIP will be used to assess pyloric diameter and distensibility, prior to and after G-POEM, performed by an endoscopist skilled in this technique. After the procedure, the patient will be observed in the hospital for 2 days. Patients will undergo an upper GI series the next day to rule out perforation. If the patient develops a complication from the procedure, he or she will be managed per standard clinical practice by the treating (unblinded) endoscopist.
  Arms: G-POEM
Procedure: Sham Gastric peroral endoscopic myotomy. — Patients assigned to the sham procedure will be treated identically as above, except for the performance of the G-POEM. Endoscopy and EndoFLIP will be performed and sedation will be stopped when the upper endoscopy is completed. Since sham endoscopy is expected to take less time than G-POEM, the patient should remain in the endoscopy procedure room for a minimum of 30 minutes (including the time required to complete the upper endoscopy). After the procedure, the patient will be observed in the hospital for 2 days. All patients will undergo an upper GI series radiographic examination the next day to rule out perforation in order to maintain study blind.
  Arms: Sham procedure

SUMMARY:
The purpose of this research is to evaluate the 12-month treatment effect of peroral endoscopic pyloromyotomy (G-POEM) vs. sham surgery in patients with gastroparesis that is not helped by medications and to analyze factors that may predict the outcome of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of chronic nausea or vomiting compatible with gastroparesis (idiopathic or diabetic) must be present for at least one year (does not have to be contiguous) prior to registration.
* Must have a mean total Gastroparesis Cardinal Symptom Index (GCSI) score of ≥ 3 at screening visit.
* Refractory gastroparesis, defined using our previously published data5, as a failure to improve over the last 6 months, despite an adequate trial of one or more standard prokinetics (metoclopramide, erythromycin, prucalopride), antinauseants (5-HT3 antagonists, promethazine, prochlorperazine, dronabinol), or neuromodulators (mirtazapine, buspirone).
* Moderate to severe delay in gastric emptying, defined as > 25% solid retained at 4 hours or > 75% retained at 2 hours. The qualifying gastric emptying scintigraphy must be performed within 18 months prior to registration or can be the baseline gastric emptying.
* No evidence of mechanical obstruction based on upper GI endoscopy or upper GI series in their medical history.

Exclusion Criteria:

* Another active disorder which could explain symptoms in the opinion of the investigator.
* Gastric retention of solids at 4 hours < 25% or < 75% at 2 hours.
* Ongoing use of prokinetic agents (e.g., metoclopramide, erythromycin, prucalopride) GLP -1 analog or agonists, or drugs that slow down gastric emptying (narcotics). Neuromodulators such as tricyclic antidepressants (amitriptyline or nortriptyline) or others that are being used at stable doses for a month prior to randomization may continue at the discretion of the care provider.
* Significant systemic illness such as chronic renal failure (adjusted for age) or liver disease as defined by Child-Pugh score of 10 or greater.
* Poorly controlled diabetes with HbA1c of greater than 10% at time of screening.
* New medications for gastroparesis-related symptoms started within 1 month prior to registration.
* Pregnancy or nursing.
* Failure to give informed consent.
* Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of the study.
* Botox injection into the pylorus within 3 months prior to registration.
* Allergy to eggs or Egg Beaters and Ensure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
GCSI-DD change | Baseline to 48 weeks post treatment
  The effect of GPOEM on nausea, early satiety, postprandial fullness, and upper abdominal pain as per changes in patient scoring in The American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index Daily Diary (ANMS GCSI-DD) which has been designed to assess symptoms associated with gastroparesis. Symptoms are rated as none (0), mild (1), moderate (2), severe (3), very severe (4) scale of the worst severity of the symptom over the last 24 hours.

SECONDARY OUTCOMES:
Change in Quality of Life as assessed by the Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life scale | Baseline to 48 weeks post treatment
  The effect of GPOEM on quality of life assessed by the Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QoL). The PAGI-QOL instrument consists of 30 items, each with response options based on a 6-point scale and with a recall period of the previous 2 weeks. The items are grouped into 5 dimensions: Daily Activities, Clothing, Diet and Food Habits, Relationship and Psychological Well-being and Distress. A score per dimension as well as a total score can be calculated. The PAGI-QOL scores range from 0 (lowest QoL) to 5 (highest QoL).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials